CLINICAL TRIAL: NCT00444808
Title: Analgesic Effect of Intranasal Calcitonin on Patients With Fractured Ribs
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Medication expired
Sponsor: Université de Montréal (Other)
Responsible Party: Raoul Daoust, University of Montreal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C.E. 2004-11-77
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Rib Fractures; Pain
Keywords: Rib fracture; Pain; intranasal calcitonin
MeSH Terms: conditions — Rib Fractures; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Intranasal calcitonin

SUMMARY:
This study, which will be conducted at the emergency room of the Sacré-Cœur hospital, requires the recruitment of 60 subjects and involves some telephone follow-up.

Calcitonin administered as an intranasal spray is already used to relieve pain caused by broken vertebrae and we seek to determine if it can be as efficient in the case of pain caused by broken ribs.This study aims at testing the hypothesis that subjects suffering from the accidental fracture of one or more ribs will get relief through the intranasal spraying of calcitonin and/or will use less opiate medication for pain relief (a combination of oxycodone chlorhydrate and acetaminophen called Percocet®).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or more.
* Accidental rib fracture (one or more) visible on a lung\thorax radiography, or on a CT Scan of the thorax, as determined by the emergency physician or the radiologist.
* The rib fracture is the main cause of pain.
* The patient says yes to the question "do you wish something for your pain" (the result of the quantitative assessment of the pain in not taken into consideration) or the patient has already received an analgesic before the initial assessment by the emergency physician.
* The patient is seen no more than 48 hours after the accident.

Exclusion Criteria:

* The patient is already receiving SC.
* Allergy or intolerance to SC, oxycodone chlorhydrate or acetaminophen
* Active neoplasia history for at least 5 years
* Toxicomania history as revealed by case history
* Osteoporosis linked to hyperparathyroidism
* Patient already using opiate analgesics or other analgesics on a regular basis (excluding aspirin at doses of 325 mg or less, as a prophylactic for cardiovascular diseases and under stable posology for at least 15 days)
* Steroid use within the past month
* Pregnancy, breast feeding
* Non-availability of patient for telephone follow-ups or follow-up appointments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-02; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Reduction of the pain level by 30% as measured on the visual analog scale of 0-100 mm on days 1, 3, 7, 14, 21, 28.
and/or reduction the use of back-up medication on days 1, 3, 7, 14, 21, 28.

SECONDARY OUTCOMES:
Improvement in the quality of life and sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Daoust, MD, Principal Investigator — Centre de recherche hôpital du Sacré-Coeur de Montréal
Locations (1):
- Hôpital du Sacré-Coeur, Montreal, Quebec, Canada